CLINICAL TRIAL: NCT07331935
Title: Clinical and Biochemical Assessment of the Effectivness of Topical Coenzyme Q10 and Topical Curcumin in Managment of Oral Leukoplakia (A Randomized Controlled Clinical Trial)
Brief Title: Efficacy of Topical Coenzyme Q10 and Curcumin for Oral Leukoplakia Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24092025
Record Dates: First submitted 2025-12-27; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Oral Leukoplakia
MeSH Terms: conditions — Leukoplakia, Oral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical Coenzyme Q10 gel (Experimental)
  Interventions: Other: Coenzyme Q10 gel
- Topical curcumin gel (Experimental)
  Interventions: Other: Topical curcumin gel

INTERVENTIONS:
Other: Coenzyme Q10 gel — Application will be performed 2-3 times daily for 4 weeks.
  Arms: Topical Coenzyme Q10 gel
Other: Topical curcumin gel — Application will be performed 2-3 times daily for 4 weeks.
  Arms: Topical curcumin gel

SUMMARY:
Oral leukoplakia (OL) is recognized as the most common potentially malignant disorder of the oral mucosa. The pathogenesis of OL is complex and multifactorial, with oxidative stress playing a central role. Topical antioxidants have gained attention as therapeutic options to help stabilize lesions and potentially prevent malignant transformation. Both CoQ10 and curcumin have demonstrated a clinical success as strong antioxidants showing their capacity to reduce the lesion size and to stabilize the disease, ultimately preventing progression into oral malignancy. Aim: This study aims to clinically and biochemically assess the effectiveness of topical Coenzyme Q10 and Curcumin in the management of homogeneous oral leukoplakia.

ELIGIBILITY:
Inclusion Criteria:

* Clinically and histologically diagnosed with homogeneous oral leukoplakia not indicated for surgical excision .
* Lesions accessible for topical application.
* Willing to sign informed consent and comply with study instructions and return to follow up

Exclusion Criteria:

* Moderate-to-severe dysplasia, carcinoma in situ, or invasive oral cancer.
* Presence of any visible oral lesions except for oral leukoplakia.
* Active periodontal diseases as this can confound salivary biomarkers.
* Significant systemic illness or immunosuppression.
* Patients who have taken systemic or topical antioxidant supplements within the last four weeks will be excluded to avoid confounding effects on salivary biomarkers.
* Pregnant and lactating women will be excluded due to hormonal changes that may alter oxidative stress and ethical considerations.
* Patients unwilling or unable to comply with study requirements.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in lesion size | baseline, 4 weeks, and 12 weeks
  measured clinically with a periodontal probe and/or digital images

SECONDARY OUTCOMES:
Change in salivary markers | baseline, 4 weeks, and 12 weeks
  Unstimulated whole saliva will be collected to assess salivary oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral medicine Department, Faculty of Dentistry, Alexandria University, Egypt, Alexandria, Egypt